CLINICAL TRIAL: NCT00925782
Title: AA Phase IIA Open-Label, Randomized, PK Comparative, Cross-Over Study of Melphalan HCL for Injection (Propylene Glycol-Free) and Alkeran for Injection for Myeloablative Conditioning in MM Patients Undergoing Autologous Transplantation
Brief Title: PK Study of Melphalan HCL & Alkeran for Injection of MA Conditioning in MM Patients of Autologous Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Acrotech Biopharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CDX-353-001
Record Dates: First submitted 2009-06-18; First posted 2009-06-22 (Estimated); Results first posted 2014-08-20 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: Multiple Myeloma
Keywords: autologous stem cell transplantation
MeSH Terms: conditions — Multiple Myeloma | interventions — Melphalan; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Melphalan-Alkeran (Other): Subjects begin with treatment Melphalan and crossover to treatment Alkeran
  Interventions: Drug: Melphalan HCL for Injection (Propylene Glycol-Free)/Alkeran for Injection; Drug: Alkeran for Injection/Melphalan HCL for Injection (Propylene Glycol-Free)
- Alkeran-Melphalan (Other): Subjects begin with treatment Alkeran and crossover to treatment Melphalan.
  Interventions: Drug: Melphalan HCL for Injection (Propylene Glycol-Free)/Alkeran for Injection; Drug: Alkeran for Injection/Melphalan HCL for Injection (Propylene Glycol-Free)

INTERVENTIONS:
Drug: Melphalan HCL for Injection (Propylene Glycol-Free)/Alkeran for Injection — Patients will be randomized to receive 100 mg/m2 of Melphalan HCL for Injection (Propylene Glycol-Free) on Day -3 and Alkeran for Injection on Day -2 prior to ASCT.
  Other Names: Evomela
Drug: Alkeran for Injection/Melphalan HCL for Injection (Propylene Glycol-Free) — Patients will be randomized to receive 100 mg/m2 of Alkeran for Injection on Day -3 and Melphalan HCL for Injection (Propylene Glycol-Free)on Day -2 prior to ASCT.
  Other Names: L-PAM, L-Sarcolysin

SUMMARY:
To assess and compare the pharmacokinetics of Melphalan HCL for Injection (Propylene Glycol-Free) versus Alkeran for Injection in multiple myeloma (MM) patients undergoing autologous stem cell transplant (ASCT).

DETAILED DESCRIPTION:
This study will be a multicenter, open-label, randomized, comparative, cross-over study of high-dose Melphalan HCl for Injection (Propylene Glycol-Free) and Alkeran for Injection conducted in 24 patients who have symptomatic MM and qualify for ASCT.

During the Study Period, patients will be randomized to receive 100mg/m2 of either Melphalan HCl for Injection (Propylene Glycol-Free) or Alkeran for Injection on Day -3 and the alternate drug product on Day -2. Blood samples for pharmacokinetic (PK) evaluation will be withdrawn through an indwelling i.v. cannula each day of melphalan dosing (Day -3 and Day -2).

Following one day of rest after the myeloablative conditioning (Day -1), patients will receive an autologous graft.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic MM requiring treatment at diagnosis or anytime thereafter.
* Patients with MM who qualify for ASCT therapy who have received appropriate primary induction therapy for transplantation.
* Adult patients (≥ 18 years old) who are 70 years of age or younger at time of transplant; patients greater than 70 years of age may qualify on a case-by-case basis if the patient meets local institutional criteria to receive a total melphalan dose of 200 mg/m2 as a conditioning regimen and if approved by the Medical Monitor.
* Patients with an adequate autologous graft which is defined as an unmanipulated, cryopreserved, peripheral blood stem cell graft containing at least 2 × 106 CD34+ cells/kg based upon patient weight.
* Patients with adequate organ function as measured by:

  * Cardiac: Left ventricular ejection fraction at rest >40% (documented within 12 weeks prior to Day -3).
  * Hepatic: Bilirubin <2 × the upper limit of normal (ULN) and ALT/AST <3 × ULN.
  * Renal: Creatinine clearance >40 mL/minutes (measured or calculated/estimated).
  * Pulmonary: DLCO, FEV1, FVC >50% of predicted value (corrected for Hgb) or O2 saturation > 92% on room air (documented within 12 weeks prior to Day -3)

Exclusion Criteria:

* Patients who have never advanced beyond Stage 1 MM since diagnosis.
* Patients who have previously received more than one autologous stem cell transplant.
* Patients with plasma cell leukemia.
* Patients with MM and systemic AL amyloidosis.
* ECOG performance status ≥2.
* Patients with uncontrolled hypertension.
* Patients with an active bacterial, viral, or fungal infection.
* Patients with prior malignancies except resected basal cell carcinoma or treated cervical carcinoma in situ. Cancer treated with curative intent >5 years previously will be allowed. Cancer treated with curative intent <5 years previously will not be allowed unless approved by the medical monitor.
* Female patients who are pregnant (positive ß-HCG) or breastfeeding.
* Female patients of childbearing potential who are unwilling to use adequate contraceptive techniques during and for 1 month following study treatment with Melphalan HCl for Injection (Propylene Glycol-Free).
* Patients seropositive for HIV.
* Patients who are unwilling to provide informed consent.
* Patients receiving other concurrent anticancer therapy (including chemotherapy, radiation, hormonal treatment, or immunotherapy, but excluding corticosteroids) within 21 days prior to the ASCT, or planning to receive any of these treatments prior to study discharge.
* Patients concurrently participating in any other clinical study.
* Patients who are hypersensitive or intolerant to any component of the study drug formulation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-01; Primary Completion 2011-06 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Omar Aljitawi, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center/University of Kansas Cancer Center and Medical Pavillion, Kansas City, Kansas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at a single study center (University of Kansas Medical Center -two facilities) in the United States under the direction of the investigator, Omar S. Aljitawi, M.D.
Pre-assignment Details: No patients that were enrolled in the study were excluded from the trial prior to assignment to groups.
Groups:
- Melphalan - Alkeran: Randomized group of Melphalan - Alkeran sequence Melphalan HCl for Injection (Propylene Glycol-Free) (single-use glass vial containing melphalan HCl 56 mg powder [equivalent to 50 mg of melphalan free base] and 2700 mg sulfobutylether-beta-cyclodextrin Captisol) reconstituted with normal saline solution, 100 mg/m2 melphalan HCl diluted with normal saline to concentration no greater than 0.45 mg/mL, infused over 30 minutes via a central venous catheter.
  Alkeran for Injection (single-use glass vial containing melphalan HCl powder [equivalent to 50 mg melphalan] and 20 mg povidone) reconstituted with sterile diluent (containing sodium citrate, propylene glycol, ethanol, and Water for Injection), 100 mg/m2 melphalan HCl diluted with normal saline to concentration no greater than 0.45 mg/mL, infused over 30 minutes via a central venous catheter.
- Alkeran - Melphalan: Randomized group of Alkeran-Melphalan
  Alkeran for Injection (single-use glass vial containing melphalan HCl powder [equivalent to 50 mg melphalan] and 20 mg povidone) reconstituted with sterile diluent (containing sodium citrate, propylene glycol, ethanol, and Water for Injection), 100 mg/m2 melphalan HCl diluted with normal saline to concentration no greater than 0.45 mg/mL, infused over 30 minutes via a central venous catheter.
  Melphalan HCl for Injection (Propylene Glycol-Free) (single-use glass vial containing melphalan HCl 56 mg powder [equivalent to 50 mg of melphalan free base] and 2700 mg sulfobutylether-beta-cyclodextrin Captisol) reconstituted with normal saline solution, 100 mg/m2 melphalan HCl diluted with normal saline to concentration no greater than 0.45 mg/mL, infused over 30 minutes via a central venous catheter.
Period: Pretreatment (Day -30 to Day -3)
Arm/Group | Melphalan - Alkeran | Alkeran - Melphalan
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0
Period: Study Period (Day -3 to Day 0)
Arm/Group | Melphalan - Alkeran | Alkeran - Melphalan
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0
Period: Follow-up(Day +1 to Date of Engraftment)
Arm/Group | Melphalan - Alkeran | Alkeran - Melphalan
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Open-label, randomized, cross-over design study where Propylene Glycol Free Melphalan and Alkeran were assessed in the same multiple myeloma patients
Arm/Group | All Study Participants
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 23
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 13
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve (0-t)
Description: AUC (0-t) was one of the pharmacokinetic endpoints to confirm pharmacokinetic similarity between Melphalan HCl for Injection (Propylene Glycol-Free) and Alkeran for Injection in patients with multiple myeloma. Pharmacokinetic similarity was defined as a difference of 20% or less in the 90% confidence intervals (CIs) for the ratios of the pharmacokinetic parameters (calculated using log-transformed data) for the two formulations.
  The AUC results provided is the summary of Melphalan PK following Melphalan-Alkeran injection in Sequence 1 and Alkeran-melphalan injection in Sequence 2.
Time Frame: Day -3 and Day -2
Population: The pharmacokinetic-evaluable population was defined as all patients who completed dosing and adequate pharmacokinetic blood draws for the calculation of AUC and Cmax for both Melphalan HCl for Injection and Alkeran for Injection.
  The results are presented by each drug group that combines data from both sequence.
Measure: Geometric Mean (Standard Deviation); unit: min*ng/mL
Groups:
- Melphalan: Open-label, randomized, cross-over design study where Propylene Glycol Free Melphalan and Alkeran were assessed in the same multiple myeloma patients. This group includes all patients with Melphalan dose administration regardless of cross over sequence
- Alkeran: Open-label, randomized, cross-over design study where Propylene Glycol Free Melphalan and Alkeran were assessed in the same multiple myeloma patients. This group includes all patients with Alkeran dose administration regardless of cross over sequence
Arm/Group | Melphalan | Alkeran
Number analyzed (Participants) | 24 | 24
min*ng/mL | 376577 (93401) [105 to 118] | 341183 (91349)

2. Secondary Outcome: Determination of Myeloablation Following Melphalan-alkeran Sequence and Alkeran-melphalan Sequence Followed by ASCT
Description: ANC <0.5 × 109/L, absolute lymphocyte count (ALC) <0.1 × 109/L, platelet count <20,000/mm3, or bleeding requiring transfusion. The first of 2 consecutive days for which cell counts drop below these cutoff levels was recorded as the date of myeloablation.
  Since the two treatments were administered consecutively with 1 day rest, the time to myeloablation and myeloablation rate was measured after both treatments were administered.
  Comparison of sequence effect was not planned in the study and due to small sample size, it was not performed.
Time Frame: 30 days
Population: The intent-to-treat (ITT) population was defined as all patients who received at least one dose of Melphalan HCl for Injection (Propylene Glycol-Free) or Alkeran for Injection. All efficacy analyses were to be performed on the ITT population.
Measure: Mean (Standard Deviation); unit: days
Groups:
- Open-label, Randomized, Cross-over Study: Open-label, randomized, cross-over design study where Propylene Glycol Free Melphalan and Alkeran were assessed in the same multiple myeloma patients
Arm/Group | Open-label, Randomized, Cross-over Study
Number analyzed (Participants) | 24
days | 3 (1)

3. Secondary Outcome: Determination of Engraftment Following Melphalan-alkeran Sequence and Alkeran-melphalan Sequence Followed by ASCT
Description: Neutrophil engraftment was defined as the first day of 3 consecutive days where ANC (absolute neutrophil count) was higher than 500/ul. The two drug treatments in this cross-over design were administered on 2 subsequent days (Day -3 and Day -2). No per arm analysis was performed.
  Since the two treatments were administered consecutively with 1 day rest, the time to engraftment and engraftment rate was measured after both treatments were administered.
Time Frame: 30 days
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Groups:
- Open-label, Randomized, Crossover Study: Open-label, randomized, cross-over design study where Propylene Glycol Free Melphalan and Alkeran were assessed in the same multiple myeloma patients undergoing transplantation.
Arm/Group | Open-label, Randomized, Crossover Study
Number analyzed (Participants) | 24
days | 11 (1)

4. Primary Outcome: Concentration-Max (Cmax)
Description: Cmax was one of the pharmacokinetic endpoints to confirm pharmacokinetic similarity between Melphalan HCl for Injection (Propylene Glycol-Free) and Alkeran for Injection in patients with multiple myeloma. Pharmacokinetic similarity was defined as a difference of 20% or less in the 90% confidence intervals (CIs) for the ratios of the pharmacokinetic parameters (calculated using log-transformed data) for the two formulations.
  The Cmax results provided is the summary of Melphalan PK following Melphalan-Alkeran injection in Sequence 1 and Alkeran-melphalan injection in Sequence 2.
Time Frame: Day -3 and Day -2
Population: The pharmacokinetic-evaluable population was defined as all patients who completed dosing and adequate subsequent pharmacokinetic blood draws for the calculation of area under the plasma concentration-time curve (AUC) and maximum plasma concentration (Cmax) for both Melphalan HCl for Injection and Alkeran for Injection.
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Melphalan | Alkeran
Number analyzed (Participants) | 24 | 24
ng/mL | 4374 (1050) [105 to 117] | 3931 (1034)

ADVERSE EVENTS:
Time Frame: Day -30 to 7 days post day of engraftment.
Description: The time between randomized sequence of treatment (24 hours) is not sufficiently long to evaluate adverse events by intervention and Adverse Events were not collected per sequence
Groups:
- All Study Participants: Open-label, randomized, cross-over design study where Propylene Glycol Free Melphalan and Alkeran were assessed in the same multiple myeloma patients undergoing transplantation. The time between randomized sequence of treatment is not sufficiently long to evaluate adverse events by intervention of or by sequence.
Arm/Group | All Study Participants
Serious Adverse Events (participants affected / at risk) | 7/24
Other Adverse Events (participants affected / at risk) | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Study Participants (N=24)
Mucosal inflammation (grade 3) (General disorders) | 2 (2)
Fatigue (grade 3) (General disorders) | 1 (1)
Febrile neutropenia (grade 3) (Blood and lymphatic system disorders) | 2 (2)
Bundle branch block (grade 3) (Cardiac disorders) | 1 (1)
Sepsis (grade 4) (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Study Participants (N=24)
Nausea (Gastrointestinal disorders) | 24 (24)
Diarrhoea (Gastrointestinal disorders) | 23 (23)
Vomiting (Gastrointestinal disorders) | 21 (21)
Dry mouth (Gastrointestinal disorders) | 11 (11)
Stomatitis (General disorders) | 9 (9)
Constipation (Gastrointestinal disorders) | 8 (8)
Abdominal pain (Gastrointestinal disorders) | 7 (7)
Dysphagia (Gastrointestinal disorders) | 6 (6)
Dyspepsia (Gastrointestinal disorders) | 3 (3)
Gastroesophageal reflux (Gastrointestinal disorders) | 3 (3)
Abdominal tenderness (Gastrointestinal disorders) | 2 (2)
Anorectal discomfort (Gastrointestinal disorders) | 2 (2)
Epigastric discomfort (Gastrointestinal disorders) | 2 (2)
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 2 (2)
Odynophagia (Gastrointestinal disorders) | 2 (2)
Oesophageal pain (Gastrointestinal disorders) | 2 (2)
Oesophagitis (Gastrointestinal disorders) | 2 (2)
Oral disorder (Gastrointestinal disorders) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 21 (21)
Decreased appetite (Metabolism and nutrition disorders) | 15 (15)
Fluid retention (Metabolism and nutrition disorders) | 10 (10)
Dehydration (Metabolism and nutrition disorders) | 5 (5)
Hyponatraemia (Metabolism and nutrition disorders) | 4 (4)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (2)
Hypophagia (Metabolism and nutrition disorders) | 2 (2)
Hypophosphataemia (Metabolism and nutrition disorders) | 2 (2)
Fatigue (General disorders) | 20 (20)
Mucosal inflammation (General disorders) | 11 (11)
Oedema peripheral (General disorders) | 11 (11)
Pyrexia (General disorders) | 11 (11)
Asthenia (General disorders) | 6 (6)
Chest pain (General disorders) | 5 (5)
Malaise (General disorders) | 5 (5)
Chills (General disorders) | 3 (3)
Platelet count decreased (Investigations) | 12 (12)
Weight increased (Investigations) | 9 (9)
Weight decreased (Investigations) | 4 (4)
Blood pressure increased (Investigations) | 3 (3)
White blood cell count decreased (Investigations) | 3 (3)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 9 (9)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Increased viscosity of bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dizziness (Nervous system disorders) | 15 (15)
Headache (Nervous system disorders) | 9 (9)
Hypogeusia (Nervous system disorders) | 5 (5)
Dysgeusia (Nervous system disorders) | 4 (4)
Somnolence (Nervous system disorders) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 (3)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 7 (7)
Thrombocytopenia (Blood and lymphatic system disorders) | 7 (7)
Febrile neutropenia (Blood and lymphatic system disorders) | 6 (6)
Rash (Skin and subcutaneous tissue disorders) | 4 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3)
Petechiae (Skin and subcutaneous tissue disorders) | 3 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Tachycardia (Cardiac disorders) | 5 (5)
Sinus tachycardia (Cardiac disorders) | 4 (4)
Hypotension (Vascular disorders) | 6 (6)
Orthostatic hypotension (Vascular disorders) | 3 (3)
Pollakiuria (Renal and urinary disorders) | 3 (3)
Vision blurred (Eye disorders) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution/PI shall submit to the Sponsor for comment, any manuscript or public release of information at least 90 days prior to its submission or release. If the Sponsor requires additional time in order to protect the results of the Study by patenting or otherwise, Institution agrees to delay submitting the Publication to any third party for up to an additional 90 days after the request by Sponsor. Such request, however, must be received by Institution during the 90-day review period.